CLINICAL TRIAL: NCT07191808
Title: EXPLORING EFFECTIVENESS OF LOW LEVEL LASER THERAPY IN THE TREATMENT OF PATIENTS WITH BELLS PALSY
Acronym: bells palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Shahid Ahmed, Shahid Ahmed, University of Lahore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UoL
Record Dates: First submitted 2025-07-22; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Bell Palsy; Bell's Palsy
Keywords: LLLT; Photmodulation; Low Leel LASER Thrapy; Idiopathic; 7th Nerve Palsy; Pakistan; Bells's Palsy; Bell's
MeSH Terms: conditions — Bell Palsy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be designed to assess the efficacy of Low-Level Laser Therapy in comparison to EMS treatment for patients diagnosed with idiopathic Bell's palsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low level LASER (Other): for neuroplasticity
  Interventions: Other: Low Level Laser Therapy

INTERVENTIONS:
Other: Low Level Laser Therapy — cluster method

SUMMARY:
The aim of the proposed research is to explore effectiveness of Low Level LASER Therapy in the country and to compare its effectiveness with routine physiotherapy. The societal benefit of submitted research is to formulate a guideline for physical therapy clinicians of the country to treat patients with Bell's Palsy through modern tool of Low Level LASER Therapy if found effective for improvement in quality of lives

DETAILED DESCRIPTION:
Annually, incidence of Bell's Palsy ranges between 1 to 4 per 10,000 individuals globally. From Pakistan figures highlight that the incidence rate of Bell's palsy in Pakistan may be above the international average, with many patients reporting a decline in their quality-of-life post diagnosis.

Low-Level Laser Therapy (LLLT), a modality known as photobiomodulation, has woven its way through various medical settings over the past decades. It has found applications in promoting wound healing, alleviating musculoskeletal pain, and now is being explored in the realm of neurological recovery. This non-invasive therapeutic technique employs non-thermal lasers or LEDs, aiming to stimulate and enhance the functions of our cellular machinery.

Globally Studies have proved effectiveness of Low Level LASER therapy in Bell's Palsy, with reduction of recovery time, improvement of Quality of Life and Personal wellbeing of patients of Bell's Palsy. We performed a survey exploring treatment preferences of Physical Therapy Clinicians to treat patients with Bell's Palsy; result showed routine contemporary practices of physiotherapy with Low Level LASER Therapy were low as 8% professionals.

The target population in this study will be assessed with standard outcome measures including FDI, HBS, FNLT / NCS and SBFGS. Two outcome measures FDI and HBS has been translated in Urdu and Reliability Studies have also been completed with permission from the Authors. A Case Control study has also been completed considering the risk factors for patients with Bell's Palsy. A Systematic Review completed by the researcher also found the Gap to explore the effectiveness of Low Level LASER Therapy for patients with Bell's Palsy.

The aim of the proposed research is to explore effectiveness of Low Level LASER Therapy in the country and to compare its effectiveness with routine physiotherapy. The societal benefit of submitted research is to formulate a guideline for physical therapy clinicians of the country to treat patients with Bell's Palsy through modern tool of Low Level LASER Therapy if found effective for improvement in quality of lives.

ELIGIBILITY:
Inclusion Criteria:

* • A confirmed diagnosis of idiopathic facial (Bell's) palsy by a certified neurologist or Physician is required (Heckmann, Urban, Pitz, Guntinas-Lichius, & Gágyor, 2019).

  * Both male and female patients, aged between 18 and 80 years (Holland & Bernstein, 2014).
  * Symptom onset within the range of 72 hours to 7 days (Petruzzelli & Hirsch, 1991).
  * A baseline House-Brackmann score of 2 to 4 is necessary (Bylund et al., 2021).
  * Availability for the entire trial duration and all subsequent follow-up visits.
  * Absence of any prior treatments (e.g., corticosteroids) for the current Bell's palsy episode.

Exclusion Criteria:

* • Alternate diagnoses that can explain Bell's palsy (e.g., Lyme disease, Ramsay Hunt syndrome) (Crouch, Hohman, Moody, & Andaloro, 2023).

  * History of recurrent Bell's palsy episodes.
  * Presence of severe medical conditions such as uncontrolled diabetes or autoimmune disorders.
  * Pregnancy or lactation. Use of concurrent medications that could interfere with facial nerve function.
  * Exposure to LLLT in the past 3 months.
  * Active skin infections or lesions in the targeted treatment area.
  * Conditions or medications that induce photosensitivity.
  * Cognitive impairments that may interfere with comprehension or feedback about the trial.
  * Participation in another trial in the past month.
  * Traumatic, inflammatory, or infectious conditions including trauma, nerve root issues, metabolic/spinal pathologies, previous spinal surgeries, or postpartum pain due to pregnancy (Singh & Deshmukh, 2022)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann Score | 6 weeks
  This scale is recognized for its capability to grade facial nerve dysfunction levels. The primary indicator of the treatment's efficacy will be any discernible improvement or non-worsening on this scale

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr Ashfaq Ahmed, PhD, Study Director — University of Lahore
Locations (1):
- NACE, Faisalābad, Pakistan